CLINICAL TRIAL: NCT01401361
Title: Clinical Evaluation of Contact™ Therapy™ Cool Path™ Cardiac Ablation System in Conjunction With EnSite Velocity Contact™ Technology for the Treatment of Typical Atrial Flutter
Brief Title: Atrial Flutter Ablation With Contact Therapy Cool Path Ablation System Along With EnSite Velocity Contact System
Acronym: CONTACT_AFL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90064772
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Typical Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Atrial Flutter RF Ablation treatment with the Contact Therapy Cool Path ablation catheter, 1500 T9 V1.43 RF Generator, Model 1611 connection cable, EnSite Velocity Contact™ Kit, and EnSite Velocity Contact software controlled via entitlement.
  Interventions: Device: Treatment Arm

INTERVENTIONS:
Device: Treatment Arm — The investigational parts of the system consists of Contact Therapy Cool Path ablation catheter, 1500 T9 V1.43 RF Generator, Model 1611 connection cable, EnSite Velocity Contact™ Kit, and EnSite Velocity Contact software controlled via entitlement .
  Other Names: Ablation with Contact Therapy Cool Path system

SUMMARY:
To demonstrate that the use of Contact Therapy™ Cool Path™ ablation catheter in conjunction with the EnSite Velocity Contact Technology for the treatment of typical atrial flutter

* Does not result into unacceptable risk of intra-procedural composite serious adverse events and,
* Does not affect efficacy of the ablation procedure The study will also evaluate the

DETAILED DESCRIPTION:
This will be a prospective, multi-center and non-randomized study. All enrolled patients who meet the eligibility criteria will receive ablation therapy for typical atrial flutter using the Contact Therapy™ Cool Path™ Cardiac Ablation System. Historical data from published (PMA P060019 Cool Path) , reported (IDE G090109 Cool Path Duo) and published literature on Atrial Flutter RF ablation studies is used to determine performance goals for primary study endpoints and derive the sample size. In addition, the following analyses will be performed in the study

1. Validation of ECI against conventional methods of assessing tip tissue contact and
2. Ancillary analysis to assess the relationship between the ECI and study outcomes. Subjects will undergo two follow up visits at day 10 and month 3 post procedure. The following assessments will be performed during these visits:

   * ECG
   * Query regarding adverse events since the last visit
   * Assessment of anti-arrhythmic and anti-coagulation medication
   * Query regarding recurrence or repeat ablation for typical atrial flutter

ELIGIBILITY:
Inclusion Criteria:

* A signed written Informed Consent
* Presence of typical atrial flutter (cavo-tricuspid isthmus dependent)
* If subjects are receiving antiarrhythmic drug therapy (Class I or Class III AAD) for an arrhythmia other than typical atrial flutter, then they need to be controlled on their medication for at least 3 months. If a subject had typical atrial flutter before starting the AAD(s) (Class I or Class III) and then subsequently had another arrhythmia (i.e. atrial fibrillation), then the 3 month AAD criteria will not apply.
* One documented occurrence of the study arrhythmia documented by ECG, Holter, telemetry strip, or transtelephonic monitor within the past 6 months
* In good physical health
* 18 years of age or older
* Agree to comply with follow-up visits and evaluation

Exclusion Criteria:

* Prior typical atrial flutter ablation treatment
* Pregnancy
* Atypical flutter or scar flutter (non isthmus dependent)
* Significant coronary heart disease or heart failure; that is unstable angina pectoris and/or uncontrolled congestive heart failure (NYHA Class III or IV) at the time of enrollment
* A recent myocardial infarction within 3 months of the intended procedure date
* Permanent coronary sinus pacing lead
* Clinically significant tricuspid valvular disease requiring surgery and/or a prosthetic tricuspid heart valve.
* Evidence of intracardiac thrombus or a history of clotting disorders
* Participation in another investigational study
* Cardiac surgery within 1 month prior to the intended procedure date
* Allergy or contraindication to Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Chinitz, MD, Principal Investigator — NYU Langone Health
Locations (20):
- United States (19):
  - Cardiology, P.C., Birmingham, Alabama
  - Aurora Denver Cardiology, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - St. Vincent's Hospital, Jacksonville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - New York University Langone Medical Center - Tisch Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Ohio Health Research Institute - GMC, Columbus, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Texas Health Research & Education Institute, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Virginia Cardiovascular Specialists, Richmond, Virginia
- Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Contact Therapy Cool Path ablation system in conjunction with EnSite Velocity Contact system : The investigational parts of the system consists of Contact Therapy Cool Path ablation catheter, 1500 T9 V1.43 RF Generator, Model 1611 connection cable, EnSite Velocity Contact™ Kit, and EnSite Velocity Contact software controlled via entitlement .
Period: Overall Study
Arm/Group | Treatment Arm
Started | 150
Completed | 122 (16 subjects were withdrawn prior to the use of the investigational device)
Not Completed | 28
Not completed — Withdrawal by Subject | 16
Not completed — Lack of Efficacy | 6
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 3
Not completed — Subject/family decision post procedure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.82 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 125
Region of Enrollment [Number; unit: participants]
  United States | 140
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety:Incidence of Composite, Serious Adverse Events Within 7 Days Post Procedure
Description: Primary safety is defined as the incidence of composite, serious adverse events within 7 days post-procedure, regardless of whether a determination can be made regarding device relatedness.
Time Frame: 7 days
Population: 150 subjects who met Inc/Excl criteria were enrolled. 16 subjects were withdrawn prior to the use of the investigational device, thus,134 were treated. 3 subjects had composite adverse events that were serious and occurred within 7 days of the ablation procedure. These events are part of the primary safety endpoint analysis per protocol.
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 134
participants | 3

2. Primary Outcome: Primary Efficacy
Description: Primary efficacy or Acute success is defined as achievement of bidirectional block in the cavo-tricuspid isthmus and non-inducibility of typical atrial flutter at least 30 minutes following the last RF ablation with the investigational system.
Time Frame: 30 minutes
Population: 134 subjects were treated with the investigational catheter and system with 1 subject failing to pass the bidirectional block inducibility test 30 minutes post ablation. Thus 133 subjects comprised the primary efficacy cohort.
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 133
participants | 129

3. Secondary Outcome: Secondary Efficacy
Description: Secondary efficacy / Chronic success is defined as freedom from recurrence of typical atrial flutter 3 months post ablation. Flutter recurrence will be documented on an ECG (or similar such as Holter, telemetry, rhythm strips, etc.). Repeat ablations, new antiarrhythmia medication (Class Ia, Ic, or III) or increase in the dosage of existing anti-arrhythmic medication (Class 1a,
  1c, III) during the 3 months post ablation are considered chronic failures.
Time Frame: 3 months
Population: 134 subjects were treated with the investigational catheter and system with 10 subjects experiencing recurring AFL. Thus 124 subjects comprised the secondary efficacy cohort (freedom from AFL at 90 days).
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 124
participants | 110

ADVERSE EVENTS:
Description: 150 subjects who met Inc./Excl. criteria were enrolled. 16 subjects were withdrawn prior to the use of the investigational device, thus,134 received the device. 3 subjects had composite adverse events that were serious and occurred within 7 days of the ablation procedure. These events are part of the primary safety endpoint analysis per protocol.
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 3/134
Other Adverse Events (participants affected / at risk) | 10/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=134)
Congestive Heart Failure (Cardiac disorders) | 1
Intermittent High Grade AV Block (Cardiac disorders) | 1
Transient Ischemic Attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=134)
Arrhythmia (Cardiac disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other